CLINICAL TRIAL: NCT04994236
Title: Efficacy and Safety of Hepatic Artery Infusion Chemotherapy in Patients With Advanced or Unresectable Hepatocellular Carcinoma Who Have Progressed or Are Intolerant to Systemic Therapy
Brief Title: Hepatic Artery Infusion Chemotherapy for Unresectable Hepatocelluar Carcinoma Who Failed to Systemic Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hui-Chuan Sun (Other)
Responsible Party: Sponsor-Investigator, Hui-Chuan Sun, Professor of Surgery, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2LHAIC
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic artery infusion chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatic Artery Infusion Chemotherapy (Experimental): Subjects assigned to this arm will receive chemotherapy via catheterizations placed into the hepatic artery.
  Interventions: Drug: Hepatic artery infusion chemotherapy with FOLFOX regimens (oxaliplatin, fluorouracil, and leucovorin)

INTERVENTIONS:
Drug: Hepatic artery infusion chemotherapy with FOLFOX regimens (oxaliplatin, fluorouracil, and leucovorin) — The FOLFOX regiments were given via hepatic artery catheterization, including oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, fluorouracil bolus 400 mg/m2, followed by fluorouracil infusion 2400 mg/m2 for 46 hours. If no severe adverse events occurred, the treatment will be repeated every 3 weeks.
  Other Names: HAIC

SUMMARY:
There are limited treatment options for patients with unresectable hepatocellular carcinoma (HCC) who failed to the combination therapy with targeted agents plus anti-PD-1/PD-L1. Hepatic artery infusion chemotherapy (HAIC) had shown potent antitumor effects in single-centered studies when was used as first-line therapy. However, HAIC was not used as second or third-line therapy.

DETAILED DESCRIPTION:
The combination therapy of anti-angiogenic agents and anti-PD-1/PD-L1 antibodies had shown potent anti-tumor efficacy for unresectable or advanced hepatocellular carcinoma. However, the treatment options were limited when patients were failed the combination therapies. Hepatic artery infusion chemotherapy (HAIC) had shown potent anti-tumor efficacy with an acceptable safety profile as a first-line treatment for patients with intermediated-stage or advanced-stage hepatocellular carcinoma. In this study, the investigators aimed to evaluate the efficacy and safety of HAIC were used in the late-line setting, i.e., after the failure of combination therapy with anti-angiogenic agents and anti-PD-1/PD-L1 antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma diagnosed histologically/cytologically, or meeting the clinical diagnostic criteria of the "Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma (2019 Edition)."
* Unresectable or advanced hepatocellular carcinoma that was assessed by the investigator. Advanced hepatocellular carcinoma was defined as BCLC C stage or Chinese Liver Cancer stage (CNLC) IIIa or IIIb stage.
* Had at least one measurable lesion in the liver.
* Liver function Child-Pugh classification of A or B7.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Patients who have received combination therapy with targeted agents combined with immune checkpoint inhibitors and have developed intolerable adverse effects or imaging confirmed intrahepatic tumor progression and have signed an informed consent form. Targeted agents include sorafenib, lenvatinib, donafenib, regorafenib, apatinib, bevacizumab (or biosimilar), and anlotinib; immune checkpoint inhibitors (mainly PD-1/PD-L1 antibodies) include pembrolizumab, nivolumab, camrelizumab, sintilimab, toripalimab, atezolizumab, and tislelizumab. Additional eligible subjects: subjects who have received at least one HAIC treatment were entered into safety evaluation (SAS); subjects who have received at least one imaging evaluation after treatment were entered into effectiveness evaluation (ITT).
* Adequate bone marrow and organ function. Reassessment of bone marrow and organ function as described above is required prior to each HAIC treatment.

  * Leukocytes ≥ 3 x 10^9/L within the last 14 days.
  * Platelets ≥ 50×10^9/L in the last 14 days without transfusion.
  * hemoglobin ≥ 90 g/L in the last 14 days without blood transfusion or erythropoietin administration.
  * total bilirubin ≤ 2 x the upper limit of normal (ULN)
  * albumin ≥ 30 g/L in the absence of human albumin or plasma transfusion within the last 14 days
  * AST and ALT ≤ 3 x ULN.
  * serum creatinine at ≤1.5×ULN.
  * International Normalized Ratio (INR) of prothrombin time ≤ 1.5×ULN.
  * Serum HBV DNA < 2 x 10^3 IU/mL; for HBV DNA > 2 x 10^3 IU/mL, treatment with nucleoside analogs for at least 1 week.
* Without grade 3 or higher adverse events (NCI CTCAE 4.0 criteria) induced by previous systemic therapy, or grade 3 or higher events reactions have recovered to grade 2 or lower.

Exclusion Criteria:

* Pathologic diagnosed with mixed liver cancer, fibrous lamellar cell carcinoma or other non-hepatocellular malignancy component.
* Previous or concurrent other malignancies, except adequately treated non-melanotic skin cancer, carcinoma in situ of the cervix, and papillary thyroid cancer
* History of organ transplantation or hepatic encephalopathy.
* Hypersensitivity to iodine-containing contrast agents, oxaliplatin, calcium folinic acid, and fluorouracil.
* History of gastrointestinal perforation and/or fistula within 6 months, history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection complicated by chronic diarrhea), Crohn's disease, ulcerative colitis, or long-term chronic diarrhea.
* Uncontrollable hypertension, systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg after optimal medical therapy, history of hypertensive crisis or hypertensive encephalopathy.
* Gastrointestinal bleeding due to portal hypertension within 6 months; G3 varices by gastrointestinal endoscopy within 3 months.
* Subjects requesting withdrawal of informed consent.
* Other circumstances that the investigator deems inappropriate for participation in the clinical trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 49 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response of intrahepatic lesions | up to 1 year
  Subjects with complete response or partial response assessed by RECIST v1.1 criteria.

SECONDARY OUTCOMES:
duration of response of intrahepatic lesions | up to 1 year
  the interval between the time of partial or complete response to the time of progressive disease in intrahepatic lesions.
Progression free survival | up to 1 year
  the interval between the time of first HAIC treatment to the time of progressive disease or patient death
Overall survival | up to 2 year
  the interval between the time of first HAIC treatment initiation to the time of patient death
Treatment cycles of HAIC | up to 1 year
  the total cycles of HAIC treatments, when the subjects could not tolerate HAIC or lose the benefit from HAIC treatment, HAIC will be discontinued.
Ratio of R0 resection | up to 1 year
  The ratio of subjects who underwent R0 resection to subjects received who received at least 1 cycle of HAIC.
The rate of adverse events | up to 1 year
  Nature, incidence, severity and seriousness of the adverse events. Adverse events are graded according to the NCI-CTCAE (Version 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Sun, MD&PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He MK, Liang RB, Zhao Y, Xu YJ, Chen HW, Zhou YM, Lai ZC, Xu L, Wei W, Zhang YJ, Chen MS, Guo RP, Li QJ, Shi M. Lenvatinib, toripalimab, plus hepatic arterial infusion chemotherapy versus lenvatinib alone for advanced hepatocellular carcinoma. Ther Adv Med Oncol. 2021 Mar 25;13:17588359211002720. doi: 10.1177/17588359211002720. eCollection 2021. PMID 33854567
- [Background] Zhou J, Sun H, Wang Z, Cong W, Wang J, Zeng M, Zhou W, Bie P, Liu L, Wen T, Han G, Wang M, Liu R, Lu L, Ren Z, Chen M, Zeng Z, Liang P, Liang C, Chen M, Yan F, Wang W, Ji Y, Yun J, Cai D, Chen Y, Cheng W, Cheng S, Dai C, Guo W, Hua B, Huang X, Jia W, Li Y, Li Y, Liang J, Liu T, Lv G, Mao Y, Peng T, Ren W, Shi H, Shi G, Tao K, Wang W, Wang X, Wang Z, Xiang B, Xing B, Xu J, Yang J, Yang J, Yang Y, Yang Y, Ye S, Yin Z, Zhang B, Zhang B, Zhang L, Zhang S, Zhang T, Zhao Y, Zheng H, Zhu J, Zhu K, Liu R, Shi Y, Xiao Y, Dai Z, Teng G, Cai J, Wang W, Cai X, Li Q, Shen F, Qin S, Dong J, Fan J. Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma (2019 Edition). Liver Cancer. 2020 Dec;9(6):682-720. doi: 10.1159/000509424. Epub 2020 Nov 11. PMID 33442540
- [Background] Finn RS, Ikeda M, Zhu AX, Sung MW, Baron AD, Kudo M, Okusaka T, Kobayashi M, Kumada H, Kaneko S, Pracht M, Mamontov K, Meyer T, Kubota T, Dutcus CE, Saito K, Siegel AB, Dubrovsky L, Mody K, Llovet JM. Phase Ib Study of Lenvatinib Plus Pembrolizumab in Patients With Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2020 Sep 10;38(26):2960-2970. doi: 10.1200/JCO.20.00808. Epub 2020 Jul 27. PMID 32716739